CLINICAL TRIAL: NCT04656899
Title: Connected Pharmacy Platform to Improve Adherence to Buprenorphine- Naloxone Prescription Treatment of Opioid Use Disorder.
Brief Title: Mobile Medication Adherence Platform for Buprenorphine-Naloxone During Treatment of Opioid Use Disorder: Phase I Study
Acronym: MAP4BUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sterling McPherson, Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB 17809; 1R44DA049629-01 (NIH)
Record Dates: First submitted 2020-09-15; First posted 2020-12-07 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pillsy arm (Active Comparator): Participants in the Pillsy arm will receive a prescription for buprenorphine-naloxone with an ''active'' Pillsy smart cap that will continuously collect data on pill bottle openings, missed doses, text messages sent, automated phone calls made. A participant who misses an entire day of buprenorphine-naloxone will automatically receive a survey about cravings and risk of relapse.
  Interventions: Behavioral: Reminders messages to improve adherence.
- Service as usual arm (No Intervention): Participants in the Service As Usual arm will receive a prescription for buprenorphine-naloxone with an ''inactive'' Pillsy smart cap that will track openings but will not provide reminders or any other messaging. They will receive a basic application that can deploy patient satisfaction surveys.

INTERVENTIONS:
Behavioral: Reminders messages to improve adherence. — If the participant does not take their medicine at the correct time, a light on the smart pill cap begins to flash. If the bottle is not opened within 20 minutes, the Pillsy application sends an SMS text reminder to the participant's phone. If the bottle is not opened within 60 minutes, the participant receives an automated phone call. The participant may also receive brief motivational phrases or craving surveys that can be tailored to participant needs and preferences. Also, based on pre-populated and adjustable craving and withdrawal levels, the participants' provider could be contacted automatically based on the thresholds being crossed. Pillsy also includes a "Pillsy Helpers" feature in which the patient can name friends and family members who will also receive a text message notification one hour after a missed dose.
  Other Names: Flashing cap; Automated phone call.
  Arms: Pillsy arm

SUMMARY:
The investigators will conduct a phase I study involving 41 participants selected randomly among patients prescribed buprenorphine-naloxone for opioid misuse as a feasibility trial of the study of the Pillsy device. The study will track the effectiveness of the Pillsy technology and associated smartphone application by measuring adherence to buprenorphine-naloxone therapy and patient satisfaction with the application and the Pillsy device.

DETAILED DESCRIPTION:
The purpose of this randomized, controlled trial in Phase I is to determine whether the Pillsy intervention can improve adherence to buprenorphine-naloxone compared to Service As Usual.

This will be a collaborative study between WSU, Pillsy, Inc, and the clinical site Ideal Options (opioid use and other substance use disorders treatment center). The overarching goal is to evaluate if the use of the Pillsy system will improve treatment adherence. The study coordinator will work closely with the clinical site, conducting a scripted screening, by phone or in person, documenting substance use, addiction treatment history, medical and psychiatric history, medication, addiction treatment goals, and availability of social support.

The Pillsy device is a smart cap that tracks pill bottle openings and uses lighted reminders to prompt patients when to take their medication. The Pillsy Helper feature is a smartphone application that sends text and phone reminders as well as links to the participant named family and friend support networks. The Pillsy Helpers feature allows participants to name friends and family members who will also receive a text message notification 1 hour after a missed dose to reach out to offer support. In addition, the prescriber will be contacted when the patient has missed a dose, giving the prescriber the opportunity to intervene. Study participants will be randomized to one of two groups. The control group will receive the Pillsy cap alone. The active group will receive the Pillsy cap and smartphone application with associated benefits. To measure adherence, all participants will provide a urine sample at each study visit and complete a questionnaire (ex: AUDIT, Fagerstrom, Addiction Severity Index, Timeline Follow-Back) and survey that assesses their satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject can and has signed an Institutional Review Board (IRB) approved informed consent form (ICF).
* Age ≥18 and ≤60 years.
* Meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnostic criteria for Opioid use disorder (OUD).
* In the professional opinion of the prescribing provider, the patient requires buprenorphine-naloxone for Opioid use disorder.
* Owns a working smartphone.
* Agrees to abstain from opioids other than Opioid Agonist Therapy (OAT) during the study.
* Able to read and speak English.
* Can identify one study partner/caregiver who agrees to participate.

Exclusion Criteria:

* Have been prescribed chronic OAT treatment in the previous 12 months.
* Have known hypersensitivity to buprenorphine and/or naloxone.
* Are pregnant or lactating women or women of childbearing potential who are not using any form of birth control.
* Have a primary diagnosis of substance use disorder other than OUD or nicotine.
* Require opioids for the treatment of chronic pain.
* Have evidence of coagulopathy within 90 days prior to enrollment.
* Have clinically significant thrombocytopenia.
* Have screening serum aspartate (AST) and alanine aminotransferase (ALT) levels 3-fold higher than upper limits of normal.
* Have screening total bilirubin or creatinine levels 1.5-fold higher than the upper limits of normal.
* Use of other medications that are known to affect the outcome measures in this study including methadone.
* Are unable to provide voluntary informed consent.
* Have pending legal issues that could adversely affect the participant's freedom to participate.
* Cannot read or speak English.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2020-12-06 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sterling McPherson, Ph.D., Principal Investigator — Washington State University; Jeffrey LeBrun, Principal Investigator — Pillsy, Inc.
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from Buprenorphine and Buprenorphine/Naloxone clinics in the NW USA region
Pre-assignment Details: 84 individuals were assessed for eligibility, of these 41 were randomized
Period: Overall Study
Arm/Group | Pillsy Arm | Service as Usual Arm
Started | 19 | 22
Completed | 16 | 13
Not Completed | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pillsy Arm | Service as Usual Arm | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (8.1) | 37.7 (11) | 36.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 7 | 12 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 2 | 0 | 2
  White | 16 | 20 | 36
  Black | 0 | 2 | 2
  Prefer not to say | 1 | 0 | 1
Employment [Count of Participants; unit: Participants]
  Unemployed | 11 | 13 | 24
  Employed | 8 | 9 | 17
Marital Status [Count of Participants; unit: Participants]
  Single | 5 | 15 | 20
  Married | 9 | 3 | 12
  Divorced | 5 | 4 | 9
Last Buprenorphine Initiation [Count of Participants; unit: Participants]
  Not Eligible | 0 | 1 | 1
  0 to 30 days ago | 5 | 8 | 13
  31 to 60 days ago | 2 | 1 | 3
  60 to 90 days ago | 2 | 1 | 3
  91 to 120 days ago | 9 | 11 | 20
  Missing | 1 | 0 | 1
Baseline Opioid Use Disorder (OUD) Diagnostic and Statistical Manual (DSM) Diagnosis [Count of Participants; unit: Participants]
  Mild | 9 | 5 | 14
  Moderate | 0 | 2 | 2
  Severe | 10 | 15 | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Medication Possession Ratio
Description: Change in adherence to buprenorphine-naloxone treatment assessed by medication possession ratio (MPR). This was calculated as mean over the course of the trial. MPR is the sum of the days' supply for all fills of a given drug in a particular time period, divided by the number of days in the time period (time period varies based on length of prescription given by provider). MPR is typically expressed as a percentage, however below we express it as the result of the fraction.
  This measurement was based on pharmacy fills (days supply).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Medication supply / days in time period
Arm/Group | Pillsy Arm | Service as Usual Arm
Number analyzed (Participants) | 19 | 22
Medication supply / days in time period | 0.839 (0.652) | 0.752 (0.713)

2. Secondary Outcome: Participant Engagement
Description: Participant engagement quantified through days of retention in treatment.
Time Frame: 12 weeks (Assessed at screening visit, week 1 visit, week 6 visit and week 12 visit)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Pillsy Arm | Service as Usual Arm
Number analyzed (Participants) | 19 | 22
Days | 71.3 (28.2) | 52.6 (38.8)

3. Secondary Outcome: Week 1, Number of Participants Satisfied With Pillsy Usability and Reminder Feedback System
Description: Week 1 "Pillsy Satisfaction Survey". "Yes" vs "No" question: "Are you satisfied with the Pillsy system overall?". Outcome data measured is count of participants endorsing yes.
Time Frame: Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pillsy Arm | Service as Usual Arm
Number analyzed (Participants) | 18 | 20
Participants | 14 | 17

4. Secondary Outcome: Number of Days Participant Self-reported Other Substance Use
Description: Participant self-report of other substance use (alcohol, cigarettes, and illicit opioids) is assessed with Timeline Follow-back measure
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Days of use
Arm/Group | Pillsy Arm | Service as Usual Arm
Number analyzed (Participants) | 19 | 22
Days of use
  Alcohol | 0.82 (3.89) | 0.24 (0.83)
  Cigarettes | 7.83 (12.81) | 9.02 (13.06)
  Illicit opioids | 0.33 (2.04) | 0.45 (2)

5. Secondary Outcome: Change in Use of Non-prescribed Opioids
Description: Use of non-prescribed opioids is assessed via urinalysis (UA) by the treatment team at Ideal Option, as a standard of care. Ideal Option will share this data with the study team (through signed data use agreement). Our study team will evaluate change in use of non-prescribed opioids over the course of the study, based on the data provided by the clinic. Below it is expressed as the mean number of illicit opioid positive UAs submitted out of the total number of UAs submitted for each arm.
Time Frame: 12 weeks
Population: Participants in both groups (Pillsy and SAU) were asked by their medical provider frequently to provide urine samples as part of their standard of care treatment. This was not on a set schedule. Results of all urinalyses were provided to the research team for analysis to evaluate change in use of non-prescribed opioids over the course of the study.
Measure: Mean (Standard Deviation); unit: Urinanalysis
Units Other Than Participants: Urinalysis
Arm/Group | Pillsy Arm | Service as Usual Arm
Number analyzed (Participants) | 19 | 22
Number analyzed (Urinalysis) | 71 | 75
Urinanalysis | 2.17 (7.25) | 1.68 (4.39)

6. Secondary Outcome: Week 6, Number of Participants Satisfied With Pillsy Usability and Reminder Feedback System
Description: Week 6 "Pillsy Satisfaction Survey". "Yes" vs "No" question: "Are you satisfied with the Pillsy system overall?" Outcome data measured is count of participants endorsing yes.
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Pillsy Arm | Service as Usual Arm
Number analyzed (Participants) | 16 | 14
Participants | 14 | 11

7. Secondary Outcome: Week 12, Number of Participants Satisfied With Pillsy Usability and Reminder Feedback System
Description: Week 12 "Pillsy Satisfaction Survey". "Yes" vs "No" question: "Are you satisfied with the Pillsy system overall?" Outcome data measured is count of participants endorsing yes.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Pillsy Arm | Service as Usual Arm
Number analyzed (Participants) | 13 | 12
Participants | 11 | 12

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Pillsy Arm | Service as Usual Arm
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/22
Other Adverse Events (participants affected / at risk) | 0/19 | 0/22

LIMITATIONS AND CAVEATS:
This was a Phase I study with the primary intention of establishing feasibility and acceptability. To determine whether or not the Pillsy intervention is effective, it is important to have a larger sample size in a Phase II trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT04656899/Prot_SAP_000.pdf